CLINICAL TRIAL: NCT00954395
Title: Optimizing the Duration of Anticoagulation in Venous Thromboembolism: the DULCIS Study
Brief Title: DULCIS (D-dimer and ULtrasonography in Combination Italian Study)
Acronym: DULCIS
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Principal Investigator, GUALTIERO PALARETI, Prof. Gualtiero Palareti, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: DULCIS
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Venous Thromboembolism
Keywords: vitamin K antagonists, D-dimer,; deep vein thrombosis, pulmonary embolism,
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism | interventions — fibrin fragment D; Fibrin Fibrinogen Degradation Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — platelet poor plasma and whole blood for Dna
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1. anticoagulation suspension: eligible patients undergo measurement of residual venous obstruction (RVO) with compression ultrasound (CUS) in case of a previous deep vein thrombosis (DVT) and/or of pulmonary artery pressure (PAP) with echocardiography in case of previous pulmonary embolism (PE). In patients with RVO is less < 4 mm in case of a previous DVT and/or PAP is normal with echocardiography in case of previous PE and in those who have undergone additional 6 months of therapy for previously altered RVO, D-dimer is measured during anticoagulation. If D-dimer is below age and gender cut-offs , anticoagulation is interrupted and D-dimer is then re-assessed after 15, 30, 60 and 90 days. If all the D-dimer measurements are below the cut-offs, anticoagulation is definitely interrupted and patients are followed-up for two years.
  Interventions: Other: D-dimer
- 2. anticoagulation prolongation: If RVO is greater than 4 mm at CUS of the lower limbs and/or PAP is increased (> 35 mmHg, > 40 mmHg in the elderly or obese), anticoagulation is prolonged for additional 6 months and the measures of RVO and/oR PAP are repeated. In those in whom PAP is altered also after 6 months of additional therapy, anticoagulation is prolonged. In patients with RVO is less < 4 mm in case of a previous DVT and/or PAP is normal with echocardiography in case of previous PE and in those who have undergone additional 6 months of therapy for previously altered RVO, D-dimer is measured during anticoagulation. If D-dimer is above age and gender cut-offs , anticoagulation is prolonged. If D-dimer is below the cut-offs , anticoagulation is interrupted and D-dimer is then re-assessed after 15, 30, 60 and 90 days. If one of these D-dimer measurement is above the cut-off , anticoagulation is resumed for at least 6 months and patients are re-evaluated.
  Interventions: Other: D-dimer

INTERVENTIONS:
Other: D-dimer — D-dimer is performed at the time of anticoagulation suspension. If above or below age and gender specific cut-offs, anticoagulation is stopped and D- dimer repeated after 15, 30, 60 and 90 days.
  Other Names: D-dimer, fibrin fibrinogen degradation products

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a standardized procedure to establish the optimal duration of anticoagulation in patients with venous thromboembolism.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE- the deposition of thrombi in the deep veins of the lower limbs-deep vein thrombosis- and/or pulmonary embolism) has an incidence of 1.0 - 1.6 events per year per 1000 persons. While the prevention and treatment of the acute phase of VTE is well established, the secondary prevention of the disease, that is its long-term management, is not well standardized. Venous thromboembolism tends to recur regardless of the duration of treatment , with an incidence of 30% over 5-10 years. Both the duration and the quality of treatment after the acute event are not well established nor consistently applied in clinical practice. Recently, the 7th Consensus Conference on Anti-thrombotic therapy of the American College of Chest Physicians recommended that patients with unprovoked VTE receive at least 3 months of anticoagulant therapy. Afterwards the risk-benefit ratio of long-term therapy should be evaluated. Long term treatment is recommended in patients at low risk of bleeding and for whom good anticoagulant monitoring is achievable. However, the risk of recurrence is greatest in the first 6 to 12 months after the initial episode while it gradually decreases thereafter. As a result, the benefits of extending anticoagulation are offset over time by the risk of clinically important bleeding associated with anticoagulation. Moreover, vitamin K antagonists (VKAs) are currently the drugs of choice, and their require a strict laboratory monitoring, but in the near future newer oral anticoagulants not requiring monitoring will be available.

Several individual characteristics such as post-anticoagulation D-dimer and residual venous obstruction have been shown to be associated with an increased risk of recurrent events. We have shown in a multicentre randomized study PROLONG (N Engl J Med 2006; 355: 1780-1789) showed that D-dimer could play a role in establishing the duration of anticoagulation after a first episode of idiopathic VTE. Patients were treated with VKA for a minimum of 3 months and D-d was tested at one month after anticoagulation withdrawal . If D-dimer was normal patients did not resume treatment, whereas those with elevated D-dimer were randomized to either stop or resume anticoagulation. Patients with an abnormal D-dimer had a statistically significant higher risk for recurrence when compared with those with normal D-d. Continued anticoagulation in patients with elevated D-d significantly reduced the risk of recurrent VTE over a follow-up of 18 months.

The purpose of this study is to evaluate the efficacy and safety of a procedure employing the evaluation of residual vein obstruction and D-dimer to establish the individual risk of recurrence and thus the necessity to prolong or stop anticoagulation ( with VKAs but also with newer anticoagulants) after venous thromboembolism.

The pre-defined objectives of the study are the following:

i) to obtain a recurrence rate < 5% per year in the first and second year after anticoagulation is suspended according to the procedure ii) to allow that after treatment for the first episode of venous thromboembolism, anticoagulation suspension in feasible in at least 40% of all subjects included in the study.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years first episode of objectively documented symptomatic idiopathic VTE, either proximal lower extremity deep vein thrombosis (DVT) and/or pulmonary embolism (PE).

Unprovoked or idiopathic , or associated with one or more of the following favouring factors

· - minor general surgery, arthroscopy or laparoscopy

* pregnancy or puerperium
* hormonal treatment (contraceptive or replacement therapy)
* travel
* minor traumas
* hospitalization in a medical ward
* reduced mobility (non complete immobilization) at least six months of VKA therapy ( or other type) for at least 3 months and not longer than 12 months ability to provide informed consent

Exclusion criteria:

* Two or more episodes of objectively documented proximal DVT and or PE ( previous distal of superficial vein thrombosis are not exclusion criteria)
* Index event was isolate distal ( calf) vein thrombosis
* Index event was PE associated with shock or prolonged hypotension at high risk
* Index event was DVT in sites different from the lower limbs
* Pregnancy or puerperium ( first 6 weeks after delivery) at the time of the visit
* Solid or haematological malignancy in the active phase or undergoing chemotherapy or radiotherapy
* Antiphospholipid antibody syndrome, diagnosed according to the Sydney criteria
* Hereditary antithrombin deficiency
* Necessity to prolong anticoagulation for any reason (due to the thrombotic event or other clinical indications
* Severe respiratory or heart failure (NYHA classes: III or IV)
* Presence of criteria indicating a short anticoagulant treatment:

Venous thromboembolism secondary to one of the following triggering factors:

* Major surgery [orthopedic, general, oncological (only if radical)]
* Bed rest (>4 dd)
* Severe trauma
* Plaster cast of the lower limbs
* high bleeding risk
* limited life expectancy,
* geographical inaccessibility
* Inability or refusal to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a first episode of venous thromboembolism attending anticoagulation clinics or general practitioners
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Recurrent venous thromboembolism (VTE) and major and minor but clinically relevant bleeding | two years after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Gualtiero Palareti, MD, Principal Investigator — St.Orsola Malpighi University Hospital
Locations (1):
- U.O. Angiologia e Malattie della Coagulazione "Marino Golinelli"; Dipartimento Cardio-Toraco-Vascolare Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

REFERENCES:
- [Background] Palareti G, Cosmi B, Legnani C, Tosetto A, Brusi C, Iorio A, Pengo V, Ghirarduzzi A, Pattacini C, Testa S, Lensing AW, Tripodi A; PROLONG Investigators. D-dimer testing to determine the duration of anticoagulation therapy. N Engl J Med. 2006 Oct 26;355(17):1780-9. doi: 10.1056/NEJMoa054444. PMID 17065639
- [Background] Legnani C, Palareti G, Cosmi B, Cini M, Tosetto A, Tripodi A; PROLONG Investigators (FCSA and Italian Federation of Thrombosis Centers). Different cut-off values of quantitative D-dimer methods to predict the risk of venous thromboembolism recurrence: a post-hoc analysis of the PROLONG study. Haematologica. 2008 Jun;93(6):900-7. doi: 10.3324/haematol.12320. Epub 2008 Apr 28. PMID 18443269
- [Background] Kearon C, Kahn SR, Agnelli G, Goldhaber S, Raskob GE, Comerota AJ. Antithrombotic therapy for venous thromboembolic disease: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):454S-545S. doi: 10.1378/chest.08-0658. PMID 18574272
- [Background] Prandoni P, Lensing AW, Prins MH, Bernardi E, Marchiori A, Bagatella P, Frulla M, Mosena L, Tormene D, Piccioli A, Simioni P, Girolami A. Residual venous thrombosis as a predictive factor of recurrent venous thromboembolism. Ann Intern Med. 2002 Dec 17;137(12):955-60. doi: 10.7326/0003-4819-137-12-200212170-00008. PMID 12484710
- [Background] Pengo V, Prandoni P. From acute pulmonary embolism to chronic thromboembolic pulmonary hypertension. Ital Heart J. 2005 Oct;6(10):830-3. PMID 16270475
- [Derived] Palareti G, Cosmi B, Antonucci E, Legnani C, Erba N, Ghirarduzzi A, Poli D, Testa S, Tosetto A, Pengo V, Prandoni P; DULCIS investigators. Duration of anticoagulation after isolated pulmonary embolism. Eur Respir J. 2016 May;47(5):1429-35. doi: 10.1183/13993003.01126-2015. Epub 2016 Feb 25. PMID 26917615
- [Derived] Palareti G, Cosmi B, Legnani C, Antonucci E, De Micheli V, Ghirarduzzi A, Poli D, Testa S, Tosetto A, Pengo V, Prandoni P; DULCIS (D-dimer and ULtrasonography in Combination Italian Study) Investigators. D-dimer to guide the duration of anticoagulation in patients with venous thromboembolism: a management study. Blood. 2014 Jul 10;124(2):196-203. doi: 10.1182/blood-2014-01-548065. Epub 2014 May 30. PMID 24879813